CLINICAL TRIAL: NCT02018042
Title: An Open-Label Single-Arm Clinical Trial to Evaluate The Efficacy of Abatacept in Moderate to Severe Patch Type Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAK2167
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; AA
MeSH Terms: conditions — Alopecia Areata | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abatacept (Experimental): Patients will be treated with abatacept 125mg subcutaneous (SC) self-administered each week. Treatment will be continued for 6 months to provide adequate time to assess the short-term efficacy and safety of abatacept in patients with alopecia areata. Patients will then be followed for an additional 6 months to assess the timing and incidence of relapse.
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — After the screening period, subjects will begin weekly self-administered subcutaneous abatacept and will continue treatment for 6 months. Patients will be instructed in self-administration of study medication at baseline (week zero) and will be observed self-administering medication at each visit. Instructions regarding study drug administration will be reinforced as needed.
  The 6-month treatment period is expected to provide adequate time to assess the short-term efficacy and safety of abatacept in patients with moderate to severe AAP. Responders will then be followed for 6 months off drug.
  Other Names: Orencia

SUMMARY:
Alopecia areata (AA) is a common disease of the immune system, known as an "autoimmune" disease. In this disease, the immune system mistakenly destroys the hair follicle, causing hair to fall out. Despite many people having this disease, research into its cause and into new, better ways to treat Alopecia Areata has lagged far behind other similar diseases of the immune system. Currently, there are no Federal Drug Administration approved drugs for Alopecia Areata.

Abatacept (made by Bristol-Myers Squibb) is a safe intervention known to effectively treat rheumatoid arthritis, another "autoimmune" disease, by fighting inflammation. There are some genetic and chemical similarities between those with active rheumatoid arthritis and Alopecia Areata, suggesting that treatment with the same drug is likely to be effective. In mice specially designed for testing drugs for the treatment of human alopecia, this medication worked to prevent the disease Alopecia Areata from starting.

To test Abatacept, we are going to treat 15 patients with moderate to severe Alopecia Areata for 6 months. Each person enrolling into this study will receive the active study drug. The effectiveness of the medication will be measured by changes in hair re-growth as determined by physical exam and photography, as well as by patient and physician scoring. Patients will be followed for another 6 months off of the drug to see if the effects of treatment last and if there is delayed response. We have recently changed the study to allow testing of abatacept in a few patients with alopecia totalis and universalis.

Small scalp biopsies and peripheral blood will be taken at the beginning of the study before treatment and then after 4,12 and 24 weeks. The chemical analysis of these skin samples and blood will help us to understand how the disease happens, how the treatment works, and perhaps even guide us to better treatments in the future.

DETAILED DESCRIPTION:
Among patients with alopecia areata, patients with higher disease burdens are unlikely to have satisfactory outcomes with current therapies. Our hypothesis is that CTLA4-Ig will be effective therapy in moderate-severe alopecia areata by blocking re-activation of CD8+ memory T cells, thereby aborting the cytotoxic T cell inflammatory response underlying alopecia areata.

Alopecia areata (AA) is a common autoimmune disease resulting from immune destruction of the hair follicle and subsequent hair loss. Despite its high prevalence, research into the pathogenesis and the development of innovative therapies in Alopecia Areata has lagged far behind other autoimmune diseases. Currently, there are no FDA approved drugs for Alopecia Areata. Abatacept is a safe intervention known to block costimulation and inflammatory responses in rheumatoid arthritis, which shares several susceptibility genes in common with Alopecia Areata. Both diseases share the involvement of CTLA4, which is the rationale for selecting Abatacept for evaluation in this clinical trial. CTLA4-Ig has been shown to prevent the onset of Alopecia Areata in the C3H-HeJ animal model of Alopecia Areata, demonstrating preclinical proof of concept data in Alopecia Areata.

We will conduct an open label pilot study of 15 patients with moderate to severe Alopecia Areata treated with SC abatacept 125mg once per week for 6 months. A few subjects with alopecia totalis or universalis will also be included. Subjects will be followed for another 6 months to evaluate durability of response following the treatment phase. The primary efficacy outcome will be the proportion of responders after 6 months of treatment compared to the historically known rate of response in untreated/placebo-treated subjects of 8 to 10%. Punch biopsies and peripheral blood will be obtained at baseline prior to treatment and then after 4, 12 and 24 weeks for immunomonitoring and molecular studies.

The safety of and incidence of adverse events related to abatacept in this population of patients will also be analyzed as a secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent Before any study procedures are performed, subjects will have the details of the study described to them, and they will be given a written informed consent document to read. Then, if subjects consent to participate in the study, they will indicate that consent by signing and dating the informed consent document in the presence of study personnel.
* Must be between 18 and 75 years of age.
* Must have a diagnosis of moderate to severe AA - defined as the presence of equal to or more than 30% and equal to or less than 95% total scalp hair loss at baseline as measured using the SALT score. In addition, a few patients with 100% scalp hair loss will be enrolled.
* Duration of hair loss must be at least 3 months.
* There may be no evidence of regrowth present at baseline.
* Subjects may be naïve to treatment or unresponsive to intralesional (IL) steroids or other treatments for AA.
* Must be willing to avoid live vaccines while on the study medication, and within 3 months of its discontinuation.
* Women of childbearing potential (WOCBP) must use highly effective methods of birth control [for up to 12 weeks after the last dose of investigational product] to minimize the risk of pregnancy]. WOCBP must follow instructions for birth control for the entire duration of the study including a minimum of 90 days after dosing has been completed.

(Acceptable methods of highly effective birth control include: Condom with spermicide, Diaphragm and spermicide, Cervical cap and spermicide)

* The use of intrauterine devices, (IUDs) shall be at the discretion of the investigator.
* Women must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of investigational product.
* Women must not be breastfeeding
* Sexually active fertile men must use highly effective birth control if their partners are WOCBP. Men that are sexually active with WOCBP must follow instructions for birth control for the entire duration of the study and a minimum of 90 days after dosing has been completed.

Exclusion Criteria:

* Sex and Reproductive Status
* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 10 weeks after the last dose of study drug.
* WOCBP using a prohibited contraceptive method.
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment or before administration of abatacept.
* Sexually active fertile men not using effective birth control if their partners are WOCBP.
* Patients with a history of or active skin disease on the scalp such as psoriasis or seborrheic dermatitis.
* Patients in whom the diagnosis of alopecia areata is in question.
* Patients with active medical conditions or malignancies (except adequately treated basal or squamous cell carcinoma) that in the opinion of the investigator would increase the risks associated with study participation, including patients with a history of recurrent infections.
* Patients with COPD
* Patients known to be HIV or hepatitis B or C positive.
* Patients with history or evidence of hematopoietic abnormality.
* Patients with history of immunosuppression or history of recurrent serious infections.
* Patients unwilling or unable to discontinue treatments known to affect hair regrowth in AA
* Coexisting disease or concurrent medications
* Patients taking TNF antagonists or other biological therapy such as anakinra.
* Patients with evidence of infection or active/untreated skin cancer.
* Patients who have been treated with intralesional steroids, systemic steroids, anthralin, squaric acid, DPCP (diphenylcycloprophenone), protopic, minoxidil or other medication which in the opinion of the investigator may affect hair regrowth within one month of the baseline visit.
* Subjects who are impaired, incapacitated, or incapable of completing study-related assessments.
* Subjects with current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, pulmonary, cardiac, neurologic, or cerebral disease, which, in the opinion of the investigator, might place a subject at unacceptable risk for participation in the study.
* Female subjects who have had a breast cancer screening that is suspicious for malignancy and in whom the possibility of malignancy cannot be reasonably excluded by additional clinical, laboratory, or other diagnostic evaluations.
* Subjects with a history of cancer in the last 5 years, other than non-melanoma skin cancers cured by local resection or carcinoma in situ. Existing non-melanoma skin cancers should be removed, the lesion site healed, and residual cancer ruled out before administration of the study drug.
* Subjects who currently abuse drugs or alcohol.
* Subjects with evidence (as assessed by the investigator) of active or latent bacterial or viral infections at the time of potential enrollment, including subjects with evidence of human immunodeficiency virus (HIV) detected during screening.
* Subjects with herpes zoster or cytomegalovirus (CMV) that resolved less than 2 months before the informed consent document was signed.
* Subjects who have received any live vaccines within 3 months of the anticipated first dose of study medication.
* Subjects with any serious bacterial infection within the last 3 months, unless treated and resolved with antibiotics, or any chronic bacterial infection (eg, chronic pyelonephritis, osteomyelitis, or bronchiectasis).
* Subjects at risk for tuberculosis (TB). Specifically excluded from this study will be subjects with a history of active TB within the last 3 years, even if it was treated; a history of active TB greater than 3 years ago, unless there is documentation that the prior anti-TB treatment was appropriate in duration and type; current clinical, radiographic, or laboratory evidence of active TB; and latent TB that was not successfully treated (≥ 4 weeks).
* Subjects known to be positive for HIV, hepatitis B or C.
* Subjects who are positive for hepatitis C antibody if the presence of hepatitis C virus was also shown with polymerase chain reaction or recombinant immunoblot assay.
* Subjects with any of the following laboratory values Hemoglobin < 10.0 g/dL WBC < 3500/mm3 (< 3 x 109/L) Platelets < 120,000/mm3 (< 3 x 109/L) Serum creatinine > 2 times the ULN Serum ALT or AST > 2 times the ULN
* Any other laboratory test results that, in the opinion of the investigator, might place a subject at unacceptable risk for participation in the study.

PROHIBITED TREATMENTS AND/OR THERAPIES:

* Subjects who have at any time received treatment with any investigational drug within 28 days (or less than 5 terminal half-lives of elimination) of the Day 1 dose.
* Any concomitant biologic DMARD, such as anakinra.
* Subjects who have been treated with intralesional steroids, systemic steroids, anthralin, squaric acid, DPCP (diphenylcycloprophenone), protopic, minoxidil or other medication which in the opinion of the investigator may affect hair regrowth within one month of the baseline visit.

OTHER EXCLUSION CRITERIA

* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-09; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Mackay-Wiggan, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center - Department of Dermatology, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biran R, Zlotogorski A, Ramot Y. The genetics of alopecia areata: new approaches, new findings, new treatments. J Dermatol Sci. 2015 Apr;78(1):11-20. doi: 10.1016/j.jdermsci.2015.01.004. Epub 2015 Jan 28. PMID 25676427

RESULTS

PARTICIPANT FLOW:
Groups:
- Abatacept: Patients will be treated with abatacept 125mg subcutaneous (SC) self-administered each week. Treatment will be continued for 6 months to provide adequate time to assess the short-term efficacy and safety of abatacept in patients with alopecia areata. Patients will then be followed for an additional 6 months to assess the timing and incidence of relapse.
  Abatacept: After the screening period, subjects will begin weekly self-administered subcutaneous abatacept and will continue treatment for 6 months. Patients will be instructed in self-administration of study medication at baseline (week zero) and will be observed self-administering medication at each visit. Instructions regarding study drug administration will be reinforced as needed.
  The 6-month treatment period is expected to provide adequate time to assess the short-term efficacy and safety of abatacept in patients with moderate to severe AAP. Responders will then be followed for 6 months off drug.
Period: Overall Study
Arm/Group | Abatacept
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Abatacept
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 39 [21 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Participants With At Least 50% Hair Regrowth
Description: The study's primary efficacy endpoint will be the proportion of responders after 6 months of treatment, with response defined as 50% or greater hair re-growth from baseline as assessed by Severity of Alopecia Tool (SALT) score at week 24. This is a relatively strict definition for defining responders and non-responders and was chosen to minimize the potential for spontaneous remission, in which fewer than 10% are expected to achieve this magnitude of hair regrowth spontaneously.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept
Number analyzed (Participants) | 15
Participants | 1

2. Secondary Outcome: Percentage of Hair Regrowth
Description: Percent hair regrowth from baseline determined by global overall improvement in SALT measurements following 24 weeks of treatment.
Time Frame: Week 24
Measure: Mean (Full Range); unit: percentage
Arm/Group | Abatacept
Number analyzed (Participants) | 15
percentage | 21.3 [2.9 to 91]

3. Secondary Outcome: Measurement of Quality of Life
Description: Quality of life measures were based on changes in the Dermatology Life Quality Index (DLQI). The DLQi is a 10-item questionnaire with each question scored from 0 (not at all) to 3 (very much). The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0 (better outcome). The higher the score, the more quality of life is impaired.
Time Frame: Baseline, Week 12, Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abatacept
Number analyzed (Participants) | 15
score on a scale
  Baseline | 4.2 (3.8)
  Week 12 | 3.9 (3.8)
  Week 24 | 4.6 (3.8)

ADVERSE EVENTS:
Time Frame: 24 weeks plus an additional 6 months post-treatment.
Description: There were no serious adverse effects, no major clinical laboratory abnormalities and no patients required discontinuation of therapy. Most common adverse event was upper respiratory infection symptoms in 6 subjects. All occurrences resolved with supportive measures and/or antibiotics. One subject experienced recurrent yeast infection. Adverse effects related to site injection was reported in 3 subjects and included body aches, tightness at the injection site, and tingling of the hands/arms.
Arm/Group | Abatacept
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 6/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept (N=15)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 6 — Upper Respiratory illnesses including common cold-like symptoms, flu, pneumonia, or otherwise associated symptoms.
Site Injection (Product Issues) | 3 — Site injection of the medication into the body included body aches, tightness at the injection site, and tingling of the hands/arms which resolved during the study period.
Candidiasis/Yeast Infection (Reproductive system and breast disorders) | 1 — Infection of the genitourinary tract which resolved with miconazole prior to the treatment end.

LIMITATIONS AND CAVEATS:
Small study size and potential for spontaneous remission that might discount the validity of clinical response. A greater observational post treatment period would strengthen conclusions. Last, inherent observer bias, by SALT scoring & photography.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT02018042/Prot_SAP_000.pdf